CLINICAL TRIAL: NCT03616509
Title: Treatment With Growth Hormone in Adults With PWS, Effect on Muscular Tone Evaluated by Functional MRI, Relationship With Strength and Body Composition
Brief Title: GH in Adults With PWS, Effect on Hypotonia Evaluated by Functional MRI, Relationship With Strength and Body Composition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Olga Gimenez-Palop, Principal Investigator, Corporacion Parc Tauli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: END-GH-2017; 2017-002164-41 (EudraCT Number)
Record Dates: First submitted 2018-07-27; First posted 2018-08-06 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Prader-Willi Syndrome
Keywords: Growth Hormone; Functional Magnetic Resonance; Strength; Body composition
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Growth Hormone

STUDY DESIGN:
Intervention Model Description: First phase: 2m with placebo Second phase: 12 m with growth hormone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Placebo and Growth Hormone (Experimental): 2 months on placebo followed by 12 months on GH
  Interventions: Drug: Growth hormone; Drug: Placebo

INTERVENTIONS:
Drug: Growth hormone — 12 months on Growth hormone, initial dose 0,2 mg per day, then adjusted by insulin like growth factor (IGF-1) level
  Other Names: Genotonorm Miniquick
Drug: Placebo — 2 months on placebo, sodium chloride 0,9% injections
  Other Names: Physiological serum (sodium chloride 0,9%)

SUMMARY:
Prader-Willi syndrome (PWS) is a genetic disorder associated with growth hormone (GH) deficiency, central hypotonia and hyperphagia that leads to life-threatening obesity. Treatment with GH in adult patients is not well stablished in guidelines of Health National System (HNS). The investigators has experience in the study of brain connectivity in these patients in relation to satiety. To date, there is no evidence about the effect of GH on central hypotonia (brain areas related with muscle tone maintenance). So, the main objective is to examine these anatomical areas before and one year after GH treatment.

Methodology: Structural and functional magnetic resonance imaging to 30 PWS patients before and after GH treatment and we will compare them to a control group.

Expected results: PWS group will show abnormal functional and structural connectivity in circuitry of muscle tone maintenance that will improve after GH treatment. These favorable changes and the absence of secondary effects will help to justify the use of this treatment and its inclusion in practical clinical guidelines of HNS for the management of this syndrome in the adulthood.

ELIGIBILITY:
Inclusion Criteria:

* PWS >=18 years with growth hormone deficit
* Signed informed consent by the patients or their legal guardian

Exclusion Criteria:

* Severe obesity
* No controled diabetes mellitus
* No treated obstructive sleep apnea or severe obstructive sleep apnea
* Active cancer
* Active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Examine brain connectivity areas related with muscle tone maintenance | 24 months
  Examine brain connectivity areas related with muscle tone maintenance making a functional MRI while the subject is making motor maneuvers, before anf after 12 months on GH treatment.

SECONDARY OUTCOMES:
Evaluation of strength | 24 months
  Evaluation of strength before and after 12 months on GH treatment
Evaluation of body composition | 24 months
  Evaluation of body composition by Dual energy x-ray absorptiometry (DEXA) before and after 12 months on GH treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olga Gimenez-Palop, MD, PhD, Principal Investigator — Corporacio Sanitària Parc Taulí
Locations (1):
- Parc Taulí Hospital Universitari, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided